CLINICAL TRIAL: NCT06849869
Title: Collaborative Care Model for Perinatal Depression Support Services -- Population-Level Equity-Centered Systems Change (COMPASS-PLUS): a Hybrid Type 2 Cluster Randomized Trial
Brief Title: Collaborative Care Model for Perinatal Wellness Support Services - Population-Level Equity-Centered Systems Change
Acronym: COMPASS+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: Brown University (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2100211; R01NR021126 (NIH)
Record Dates: First submitted 2025-02-19; First posted 2025-02-27 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-02

CONDITIONS: Perinatal Mental Health
Keywords: health services interventions; mental health; collaborative care model; compass+; perinatal care
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: randomized stepped wedge design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- COMPASS+ (Experimental): COMPASS+ services are embedded into the perinatal practice. COMPASS+ includes mental health support services and monitoring by a behavioral health care manager, a patient registry to track participant response to treatment, and weekly team huddles supervised by a perinatal psychiatrist to discussed new participants in the program or individuals who are not symptomatically improving. Patients are eligible for referral to COMPASS+ during pregnancy through one year postpartum.
  Interventions: Behavioral: COMPASS+
- Usual care (No Intervention): Perinatal care practices support the mental health needs of patients providing usual care workflows at their clinic (e.g. screening for depression and anxiety symptoms in each trimester and postpartum, referring patients to community resources)

INTERVENTIONS:
Behavioral: COMPASS+ — COMPASS+ is centered around the integration of a care manager (a licensed mental health clinician) who provides mental health supports (e.g. short-term therapy) and symptom monitoring to perinatal patients. The care manager works closely with the patient and obstetric clinician to create a treatment plan based on the patient's preferences and needs. The care manager also utilizes a care registry to send monthly mental health screeners to patients and track their symptoms. The care manger meets weekly with the obstetric clinician and a consulting psychiatrist to review and modify treatment plans as needed. The care manager services are available throughout pregnancy and up to one year postpartum.
  Arms: COMPASS+

SUMMARY:
The collaborative care model (CCM) is a health services intervention that integrates mental health care in primary care settings. The goal of this study is to adapt the CCM to the perinatal care context, including community co-designed adaptations to enhance health equity (COMPASS+). The main objectives of the study are to:

1. Evaluate the effect of COMPASS+ on depression symptom outcomes. Specifically we will evaluate population-level depression symptom trajectories and the prevalence of suicidal ideation among. We will also measure rates of depression response and remission for those who have elevated screen scores (i.e., PHQ9 ≥ 10)
2. Adapt, optimize, and evaluate COMPASS+ implementation strategies to the unique context of perinatal care and evaluate implementation outcomes. The RE-AIM framework will be used to evaluate implementation outcomes (acceptability, appropriateness, feasibility, and fidelity). We hypothesize that variability in effectiveness outcomes will be attributable to variability in fidelity to the implementation strategies or in implementation outcomes.
3. Identify the effect of COMPASS+ on perinatal depression and implementation outcomes across racial and ethnic subgroups.

DETAILED DESCRIPTION:
One in five women experiences perinatal depression (PD), defined as an episode of major depressive disorder, during pregnancy or postpartum. PD can have devastating consequences for the individual, family, and community. In its most extreme form, PD can lead directly to suicide, a leading contributor to maternal mortality (MM). Untreated PD also indirectly contributes to severe maternal morbidity (SMM) and MM via associated behavioral risk factors. Despite evidence-based recommendations for PD, only 3-5% of women with PD will achieve remission of their depressive symptoms. Gaps in addressing social determinants of mental health (SDoMH), including structural racism and discrimination, contribute to the lack of success in treating PD, particularly among pregnant and postpartum individuals. Our team has identified marked racial disparities in both screening for PD and in its actual treatment.

In contrast to the existing, but failing, systems for PD care, the collaborative care model (CCM) is an established integrated supportive care intervention built on four equity-centered core principles: 1) patient-centered team care, 2) population-based care, 3) measurement-optimized treatment, and 4) evidence-based care. In primary care settings, over 80 randomized trials have demonstrated the efficacy of the CCM for improving depression outcomes. However, CCM is not broadly utilized in obstetric care. There are two major reasons for this gap from evidence to practice. The first is the lack of rigorous and generalizable evidence to support the impact of the perinatal CCM (pCCM) on population-level depression outcomes. Second, substantive differences between obstetric and primary care, which occur at the patient, provider, and system-levels, require tailored implementation strategies for pCCM.

Our prior formative research generated an optimized package of strategies for effectively implementing pCCM within diverse perinatal care settings through COMPASS (Collaborative Care Model for Perinatal Depression Support Services). We demonstrated that COMPASS improves the steps necessary for PD care, including screening and recommending treatment for PD. Moreover, our research has demonstrated that COMPASS reduces racial disparities in the steps required for PD care. Nonetheless the small samples sizes of the available studies preclude robust analyses of impact on the racial and ethnic disparities in PD outcomes. The lack of a rigorous approach to identifying and addressing SDoMH renders even the successes of COMPASS inadequate.

The critical need to equitably and adequately care for mental health conditions in pregnancy and postpartum informs the creation of COMPASS-PLUS (Collaborative Care Model for Perinatal Depression Support Services - Population-Level Equity-Centered Systems Change) (herein referred to as COMPASS+). COMPASS+ is built upon the foundations of COMPASS and embeds an anti-racist approach to addressing SDoMH via 1) a health equity advocate and 2) race and ethnicity-centered support groups for pregnancy and postpartum people, irrespective of any identified mental health needs. We propose a multi-site hybrid type 2 implementation effectiveness stepped wedge cluster randomized trial to test our central hypothesis that COMPASS+ is more effective and equitable than standard care for PD outcomes. To test this hypothesis, six diversely structured clinics across Rhode Island will be randomized to receive COMPASS+ or usual care to address the following specific aims:

Aim 1: Evaluate the effect of COMPASS+ on depression symptom severity and rate of depression response and remission. We hypothesize that implementing COMPASS+ will improve Patient Health Questionnaire 9 (PHQ9) scores (primary outcome) and reduce suicidal ideation across the study population. We hypothesize that implementing COMPASS+ will increase depression response (50% reduction in PHQ9 compared to baseline) and depression remission (PHQ9 ≤ 9) among those with PD.

Aim 2: To adapt, optimize, and evaluate COMPASS+ implementation strategies to the unique context of perinatal care and evaluate implementation outcomes. The RE-AIM framework will be used to evaluate implementation outcomes (acceptability, appropriateness, feasibility, and fidelity). We hypothesize that variability in effectiveness outcomes will be attributable to variability in fidelity to the implementation strategies or in implementation outcomes.

Aim 3: Identify the effect of COMPASS+ on perinatal depression and implementation outcomes across racial and ethnic subgroups. We hypothesize that COMPASS+ will reduce Latinx and Black versus White disparities in COMPASS+ reach and in the aforementioned PD outcomes. A subset of women (n=30) will undergo qualitative interviews regarding their experiences with COMPASS+ to evaluate racial and ethnic differences in acceptability and accessibility, using the RE-AIM framework.

The expected outcome of this project is to generate the empiric evidence needed to understand the effect of the CCM in general, and COMPASS+ specifically, on PD-related outcomes. We will generate an optimized package of successful implementation strategies for COMPASS+ to promote broad dissemination. Findings from this trial will be broadly applicable to women throughout the United States who face challenges in receiving adequate mental health care. Moreover, our results will have a substantial impact on identifying and addressing the critical factors that contribute to racial and ethnic disparities in PD-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* all pregnant and postpartum people receiving care at participating sites
* age > 17 years

Exclusion Criteria:

* age < 18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14820 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ9) trajectories | enrollment in prenatal care through end of one year postpartum
  Depression symptom trajectories will be measured using the PHQ9
  PHQ9 scores will be collected by the perinatal practice in each trimester and again postpartum for all pregnant and postpartum people receiving prenatal care. PHQ9 scores will also be collected by the care manager every 30 days for those referred to the COMPASS+ program until one year postpartum. Each of these scores will be entered into the trajectory analysis.

SECONDARY OUTCOMES:
Suicidal ideation as assessed by the PHQ9 | enrollment in prenatal care through end of one year postpartum
  Suicidal ideation is defined as a PHQ-9 question 9 score > 0
  PHQ9 scores will be collected by the perinatal practice in each trimester and again postpartum for all pregnant and postpartum people receiving prenatal care.
  PHQ9 scores will also be collected by the care manager every 30 days for those referred to the COMPASS+ program until one year postpartum
Depression symptom response: Number of participants with a PHQ9≥10 who achieve a 50% reduction in PHQ9 | enrollment in prenatal care through end of one year postpartum
  Among participants who have an elevated screen for depression (i.e., PHQ-9≥10), the proportion of participants who achieve response (50% reduction in PHQ-9 compared to baseline) in their depression symptoms.
Depression symptom remission: Number of participants with a PHQ9≥10 who achieve a PHQ9<10 | enrollment in prenatal care through end of one year postpartum
  Among participants who have an elevated screen for depression (i.e., PHQ-9≥10), the proportion of participants who achieve remission (PHQ-9 < 10) in their depression symptoms.
Acceptability measured by the Acceptability of Intervention Measure (AIM) | early implementation (1-2 months), mid-implementation (6-7 months), and sustainment (12-13 months)
  The AIM will be completed by clinician champions and clinic stakeholders within each practice
Appropriateness measured using the Intervention Appropriateness Measure (IAM) | early implementation (1-2 months), mid-implementation (6-7 months), and sustainment (12-13 months)
  The IAM will be completed by clinician champions and clinic stakeholders within each practice
Feasibility measured using the Feasibility of Intervention Measure (FIM) | early implementation (1-2 months), mid-implementation (6-7 months), and sustainment (12-13 months)
  The FIM will be completed by clinician champions and clinic stakeholders within each practice
Maintenance measured using the Clinical Sustainability Assessment Tool (CSAT) | 12-13 months after implementation at each site
  The CSAT will be completed by the MPIs, clinician champions, and clinic stakeholders within each practice

CONTACTS AND LOCATIONS:
Locations (1):
- Women and Infants Hospital, Providence, Rhode Island, United States